CLINICAL TRIAL: NCT05276076
Title: A Prospective, Open Label, Dose-escalation, SAD/MAD, Multicenter, 24weeks, Phase I/IIa Clinical Trial to Evaluate the Safety, Tolerability and Pharmacodynamics of Investigational Product (VM-001) in Patients With Graft-versus-host Disease(GvHD)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ViGenCell Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VM-201
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part 1 Single Ascending Dose, Cohort 1 (Experimental): Cohort 1 : 1X10^6 cells/kg The safety of 2 subjects is evaluated for 1 week after single dose of IP. If CTCAE grade 3 or higher adverse drug events (ADR) do not occur in the two subjects: Begin enrollment for Cohort 2.
  Interventions: Biological: VM-001 1X10^6 cells/kg
- Part 1 Single Ascending Dose, Cohort 2 (Experimental): Cohort 2 : 3X10^6 cells/kg The safety of 2 subjects is evaluated for 1 week after single dose of IP. If CTCAE grade 3 or higher adverse drug events (ADR) do not occur in the two subjects: Begin enrollment for Cohort 3.
  Interventions: Biological: VM-001 3X10^6 cells/kg
- Part 1 Single Ascending Dose, Cohort 3 (Experimental): Cohort 3 : 5X10^6 cells/kg The safety of 2 subjects is evaluated for 1 week after single dose of IP.
  Interventions: Biological: VM-001 5X10^6 cells/kg
- Part 2 Multiple Ascending Dose, Cohort 1 (Experimental): Cohort 1 : two doses in total, 1X10^6 cells/kg per dose, weekly The safety of 3 subjects is evaluated for 4 week after two dose of IP. If CTCAE grade 3 or higher adverse drug events (ADR) do not occur in the three subjects: Begin enrollment for Cohort 2.
  Interventions: Biological: VM-001 1X10^6 cells/kg two dose
- Part 2 Multiple Ascending Dose, Cohort 2 (Experimental): Cohort 2 : four doses in total, 1X10^6 cells/kg per dose, weekly The safety of 3 subjects is evaluated for 8 week after two dose of IP.
  Interventions: Biological: VM-001 1X10^6 cells/kg four dose

INTERVENTIONS:
Biological: VM-001 1X10^6 cells/kg — Administration: Inject intravenously single dose
  Arms: Part 1 Single Ascending Dose, Cohort 1
Biological: VM-001 3X10^6 cells/kg — Administration: Inject intravenously single dose
  Arms: Part 1 Single Ascending Dose, Cohort 2
Biological: VM-001 5X10^6 cells/kg — Administration: Inject intravenously single dose
  Arms: Part 1 Single Ascending Dose, Cohort 3
Biological: VM-001 1X10^6 cells/kg two dose — Administration: Inject intravenously
  1X10^6 cells/kg per dose, two dose in total, weekly
  Arms: Part 2 Multiple Ascending Dose, Cohort 1
Biological: VM-001 1X10^6 cells/kg four dose — Administration: Inject intravenously
  1X10^6 cells/kg per dose, four dose in total, weekly
  Arms: Part 2 Multiple Ascending Dose, Cohort 2

SUMMARY:
The present study is multi center, phase I/IIa clinical trial to evaluate the safety and pharmacodynamics of investigational Product (VM-001) in patients with graft-versus-host disease(GvHD). A total of 12 subjects (Part 1 SAD[3 cohort(2 subjects/cohort)], Part 2 MAD[2 cohort(3subjects/cohort)]) are recruited.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥19 years of age
* Acute GvHD or chronic GvHD after hematopoietic stem cell transplant
* Subjects who no longer have available standard treatment.
* ANC≥1,000cells./mm^3
* AST, ALT, total bilirubin less than 3 times the upper limit of normal
* serum creatinine less than 1.5 times the upper limit of normal

Exclusion Criteria:

* Received an anti-thymocyte globulin(ATG) within 14 days before enrollment
* FCV or FEV less than 70%
* Any uncontrolled infection or active infection requiring ongoing systemic treatment
* Received an investigational agent within 6 months before enrollment.
* Evidence of bleeding diathesis or coagulopathy.
* Active hepatitis C virus (HCV) or hepatitis B virus (HBV)
* Breastfeeding or pregnant.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-11-20 (Estimated); Primary Completion 2024-11-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of VM-001 [ Time Frame: 1 week ] | 7 day cycle
  First 7-day treatment dose limiting toxicities (DLT) graded according to CTCAE in the MTD-determining population in Phase 1 based on the number of participants with adverse effects as measure of tolerability at various dose levels

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Ki Min, MD, Ph.D., Principal Investigator — The Catholic University of Korea

IPD SHARING:
Plan to Share IPD: No